CLINICAL TRIAL: NCT00491413
Title: High Dose Erythropoietin for Neonates With Asphyxia
Brief Title: Erythropoietin for Infants With Brain Injuries Due to Oxygen Deprivation at Birth
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21HD042308 (NIH)
Record Dates: First submitted 2007-06-22; First posted 2007-06-26 (Estimated); Last update posted 2007-06-26 (Estimated); Status verified 2003-08

CONDITIONS: Asphyxia
Keywords: neurodevelopmental outcomes
MeSH Terms: conditions — Asphyxia | interventions — Erythropoietin

INTERVENTIONS:
Drug: epoetin

SUMMARY:
Erythropoietin (Epo) is a hormone normally found in the body that may protect brain cells from damage due to lack of oxygen. This study will evaluate the safety of high-dose Epo in infants who did not get enough oxygen during birth.

DETAILED DESCRIPTION:
Damage to the central nervous system as a result of oxygen deprivation at birth is a major cause of life-long mental and developmental handicaps. When there is not enough oxygen in the blood (hypoxemia) the brain is deprived of oxygen. Some brain cells respond by producing Epo. Epo then binds to oxygen-deprived brain cells. This binding triggers chemical reactions within the brain cell that prevent cell death. Epo also reduces inflammation around the brain cells and acts as an antioxidant. In animal studies, recombinant Epo (rEpo) administration, even up to six hours after oxygen deprivation, reduced subsequent brain injury by 50% to 70%.

Epo has been used by neonatologists to stimulate erythropoiesis (red blood cell production) and reduce the incidence of blood transfusions. Doses of rEpo required for protection of brain cells are considerably higher than those traditionally used by neonatologists.

This study will evaluate the pharmacokinetics, biologic effect, and safety of high dose Epo in neonates with brain injury due to hypoxemia.

Within six hours of birth, each eligible infant will receive one dose of rEpo intravenously. Any infants who require a lumbar puncture during the first week of life will have levels of natural Epo and rEpo in their spinal fluid measured. Blood tests will be used to measure the antioxidant effect of Epo and the impact on red blood cell production. Neurodevelopmental outcome will be measured at 6 and 12 months of age.

ELIGIBILITY:
Inclusion Criteria

* Infant 6 hours of age or less
* Apgar scores less than or equal to 3 at 1 and 5 minutes
* Weight greater than 2500 grams (5.5 lbs)
* Central venous line in place

Exclusion Criteria

* infants are ineligible if they do not meet the inclusion criteria above

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Robert D. Christensen, MD, Principal Investigator — University of South Florida
Locations (1):
- All Children's Hospital, St. Petersburg, Florida, United States